CLINICAL TRIAL: NCT02756013
Title: A Phase II Trial of Weight-based Dosing for Dense Weekly Paclitaxel and Carboplatin in Overweight Patients With a BSA > 2.0
Brief Title: Weight-based Dosing for Dense Weekly Paclitaxel and Carboplatin in Overweight Patients w/ Body Surface Area (BSA) > 2.0
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual - terminated
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE13815
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Gynecologic Malignancies
Keywords: chemotherapy dosing; Body surface area; BSA; paclitaxel; carboplatin; dose dense
MeSH Terms: interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel + Carboplatin (Experimental): Paclitaxel dosed by actual body surface area and not maxed at BSA 2.0. The Carboplatin dose will be calculated according to the Calvert formula using as estimated glomerular filtration rate from the Cockcroft-Gault formula and will be subject to maximum allowed doses.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — 80mg/m2 IV days 1,8, and 15 every 21 days x 6-9 cycles
  Other Names: Taxol
Drug: Carboplatin — area under the curve (AUC) 6 IV day 1 every 21 days x 6-9 cycles
  Other Names: Paraplatin; Paraplatin - aqueous solution (AQ)

SUMMARY:
The purpose of this study is to evaluate the side effects and effectiveness of giving standard paclitaxel chemotherapy in doses based on actual body surface area in combination with standard dosed carboplatin chemotherapy for overweight women.

DETAILED DESCRIPTION:
Primary Objective The primary objective is to prospectively evaluate the Relative Dose Intensity (RDI) and toxicity of weight-based dose dense weekly paclitaxel and carboplatin in overweight patients with a BSA > 2.0 compared to the Japanese Gynecologic Oncology Group trial (JGOG 2016) during 6 - 9 cycles of chemotherapy.

Secondary Objective(s) The secondary objective is to evaluate progression-free survival in this patient population.

Study Design This is a descriptive study to determine what the relative dose intensity of patients who are overweight with a BSA of greater than 2.0 can achieve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed or presumed diagnosis of gynecologic malignancy for whom chemotherapy with paclitaxel and carboplatin is planned.
* Body Surface area >2.0
* Patients must have adequate:

  * Renal function: Creatinine <1.5 x Institutional upper limits of normal (ULN)
  * Bone marrow function:

    * Absolute neutrophil count (ANC) ≥ 1,500/mcl. This ANC cannot have been induced or supported by granulocyte colony stimulating factors.
    * Platelets ≥ 100,000/mcl.
  * Hepatic function:

    * Bilirubin ≤ 1.5 x ULN.
    * Aspartate aminotransferase (AST) (SGOT) ≤ 2.5 x ULN.
    * Alkaline phosphatase ≤ to 2.5 x ULN.
  * Neurologic function:

    * Neuropathy (sensory and motor) ≤ CTCAE Grade 1.
* Patients must have a Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Patients must be entered within 12 weeks of diagnosis.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients who have received prior chemotherapy.
* Patients with acute hepatitis or active infection that requires parenteral antibiotics.
* Patients with clinically significant cardiovascular disease. This includes:

  * Myocardial infarction or unstable angina < 6 months prior to registration.
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication. This does not include asymptomatic, atrial fibrillation with controlled ventricular rate.
* Patients who are pregnant or nursing.
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study.
* Patients with known allergy to cremophor or polysorbate 80.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rose, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel + Carboplatin: Paclitaxel dosed by actual body surface area (BSA) and not maxed at BSA 2.0. The Carboplatin dose will be calculated according to the Calvert formula using as estimated glomerular filtration rate from the Cockcroft-Gault formula and will be subject to maximum allowed doses.
  Paclitaxel: 80mg/m2 IV days 1,8, and 15 every 21 days x 6-9 cycles
  Carboplatin: area under the curve (AUC) 6 IV day 1 every 21 days x 6-9 cycles
Period: Overall Study
Arm/Group | Paclitaxel + Carboplatin
Started | 3
Completed | 1
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Hypersensitivity | 1

BASELINE CHARACTERISTICS:
Population: Participants who went on study
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 2
  60-69 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Relative Dose Intensity as Measured by Mean Percent of Intended Cycles Completed
Description: Prospective evaluation of the Relative Dose Intensity (RDI) of weight-based dose dense weekly paclitaxel and carboplatin as measured by the average percent of completed treatment cycles out of the intended therapeutic plan
Time Frame: Up to 190 days
Population: Participants who received treatment
Measure: Mean (Full Range); unit: percent of intended cycles completed
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 2
percent of intended cycles completed | 77.5 [66 to 89]

2. Secondary Outcome: Number of Participants With Progression-free Survival (PFS)
Description: Progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 3 months for up to 2 years, then every 6 months (up to 31 months)
Population: Participants enrolled in study. Long Term Follow Up stopped after termination of study due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 3
Participants
  3 months | 3
  6 months | 3
  9 months | 2
  12 months | 2
  15 months | 2
  18 months | 2
  21 months | 2
  24 months | 2
  31 months | 2

ADVERSE EVENTS:
Time Frame: Before each treatment, up to 189 days (21 day cycles, up to 9 cycles)
Arm/Group | Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Carboplatin (N=3)
Peripheral neuropathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02756013/Prot_SAP_002.pdf
  • Informed Consent Form (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02756013/ICF_001.pdf